CLINICAL TRIAL: NCT04349384
Title: Audit of the Quality of Surgical Treatment of Colorectal Cancer
Brief Title: Audit of Surgery for Colorectal Cancer
Acronym: AuditCR
Status: Completed | Type: Observational
Sponsor: Institut National d'Oncologie, Morocco (Other Government)
Responsible Party: Principal Investigator, Anass Majbar, Professor of surgery, Institut National d'Oncologie, Morocco
Other Study IDs: SCOD 2
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Rectal Adenocarcinoma; Colon Adenocarcinoma
Keywords: Rectal neoplasms; Colon neoplasms
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colon adenocarcinoma: Patient who underwent surgical resection for colon adenocarcinoma
  Interventions: Procedure: Colorectal resection
- Rectal adenocarcinoma: Patient who underwent surgical resection for rectal adenocarcinoma
  Interventions: Procedure: Colorectal resection

INTERVENTIONS:
Procedure: Colorectal resection — Colon or rectal resection for colorectal adenocarcinoma

SUMMARY:
The aim of this project is to audit the surgical care in patients treated for colorectal adenocarcinoma. This study focused on collecting data from all consecutive cases of colon and rectal adenocarcinoma operated at the National Institute of Oncology in Rabat during a two-years period. Using standardized forms, the investigators collected data relating to each stage of treatment: pre-therapeutic, surgical and post-operative in order to measure the quality of the surgical care delivered. These results were compared to established benchmarks and to similar audit studies carried out in other countries around the world.

DETAILED DESCRIPTION:
Quality improvement initiatives and in particular the accreditation procedure raises the inevitable question of measuring quality in health. Several surgical audits have been carried out internationally, showing the importance of collecting reliable and valid information on the quality of care. This approach allows an evaluation and improvement of the quality of care provided, significantly correlated to a direct impact on morbidity and mortality. In addition, it provides valuable information for evidence-based medicine research as it provides data on patients often excluded from therapeutic trials.

Colorectal cancer is the first digestive cancer and the third cancer worldwide. Surgical resection is the main curative treatment. Surgical quality is associated with better short and long term results. Quality improvement measures, with the goal to improve surgical care of colorectal cancer, are becoming a standard worldwide.

The aim of this project is to audit the surgical care in patients treated for colorectal adenocarcinoma. This study focused on collecting data from all consecutive cases of colon and rectal adenocarcinoma operated at the National Institute of Oncology in Rabat. Using standardized forms, the investigators collected data relating to each stage of treatment: pre-therapeutic, surgical and post-operative in order to measure the quality of the surgical care delivered. These results were compared to established benchmarks and to similar audit studies carried out in other countries around the world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven colorectal adenocarcinoma who underwent surgical resection with curative intent between 1 January 2018 and 31 December 2019.

Exclusion Criteria:

* Colon or rectal resections for other histologic types than adenocarcinoma.
* Palliative intent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients (> 18 years) who underwent surgical resection for colon or rectal adenocarcinoma, with curative intent between 1 January 2018 and 31 December 2019, at the Digestive surgical oncology department of the National Institute of Oncology in Rabat Morocco.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Retrieved lymph nodes | 1 month after surgery
  Number patients with retrieved lymph nodes after colon resection above 12
Positive circumferential margin | 1 month after surgery
  The rate of patients with circumferential margin < 1 mm on surgical specimen of rectal resection for rectal adenocarcinoma.
Morbidity | 90 days after surgery
  Morbidity assessed using using the Clavien-Dindo grading system at discharge and at 90 days after surgical resection for colorectal adenocarcinoma

SECONDARY OUTCOMES:
Pre-operative CT-scan | 7 days after surgery
  Rate of patients who had computed tomography before surgery
Multidisciplinary team meeting | 7 days after surgery
  Rate of cases who were discussed during a multidisciplinary team meeting before surgery for patients who had surgical resection for colorectal adenocarcinoma
MRI for rectal adenocarcinoma | 7 days after surgery
  Rate pf patients who had a pelvic Magnetic resonance imaging or rectal ultra-sonography in the pre-operative work-up of rectal adenocarcinoma
Anastomotic leakage | 90 days after surgery
  Rate of anastomotic leakage after resection of colorectal cancer with the creation of anastomosis
Readmission | 90 days after surgery
  Rate of hospital readmissions leakage after resection of colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Anass M Majbar, Principal Investigator — National Institute of Oncology
Locations (1):
- Institut National d'Oncologie, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided
Under reasonable request, we would share individual patient data